## A rehabilitation tool to determine patient's stay in hospital after joint replacement

Protocol director: Dr. Derek Amantullah

Study coordinator:

Introduction: SPARTA science has developed a post-operative rehab tool allowing the surgeon and the entire healthcare staff to optimize care according to the patient's specific needs. The Sparta Platform includes force plate hardware coupled with Sparta Scan software that enables quick assessment of an individual's movement and balance within minutes

The Sparta Scan takes a comprehensive look into an individual's movement qualities by measuring force production. The magnitude as well as efficiency of force production is analyzed to determine the progress of the patients on predicted trajectories of recovery, and more easily identify and triage those few patients who might have to stay longer in hospital facility.

As part of an integrated clinical care pathway, post-operative scoring of likelihood of discharge is an attractive prospect, because it allows caregivers to focus on patients who require the most assistance with obtaining safe and appropriate postoperative care.

| Purpose | To obtain an objective score which is patient-centered, datadriven, and value-based solution for post-operative rehabilitation. |
|---|---|
| Eligibilty criteria | Joint replacement surgery, age should be more than or equal to 18 years. |

NCT03777007 October 8, 2021

| Study type | Prospective observational study |
|---|---|
| Sample size | 60 |
| Endpoints | Primary endpoint: Length of stay in hospital. Higher the score, shorter is the stay. Secondary endpoint: Reliability on force plate to co-relate with clinical data on data points such as discharge location, gait aid use, Knee society score(KSS) and range of motion(ROM). Time intervals for recording Gait aid use, KSS and ROM are as - 1. Gait aid use at the time of discharge, 2 weeks follow up, 6 weeks follow up, 3 weeks follow up, 1 year follow up and 2 year follow up 2. Outcome score (KSS) at 3 weeks follow up, 1 year follow up and 2 year follow up 3. Range of motion at 2 weeks follow up, 3 months follow up, 1 year follow up, 6 weeks follow up, 1 year follow up, 6 weeks follow up, 1 year follow up, 3 months follow up, 1 year follow up and 2 year follow up |
| PROM used | KOOS JR, PROMIS & KSS |
| Budget | TBD |
| Personnel | IRB submission & data collection |
| I CISUIIICI | מאווווטטוטוז א עמנמ נטוובננוטוז |

NCT03777007 October 8, 2021

| Dr. Derek F. Amanatullah, M.D., |
|---------------------------------|
| Ph.D |
| Phone: |
| Email: dfa@stanford.edu |
| Phone : |
| Email: |

NCT03777007 October 8, 2021